CLINICAL TRIAL: NCT02262559
Title: Bioequivalence Study of BIBR 277 Tablet (Erythritol Based) Compared With Its Capsule Formation in Healthy Male Volunteers
Brief Title: Bioequivalence of BIBR 277 Tablet Compared With Capsule in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 502.414
Record Dates: First submitted 2014-10-09; First posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Telmisartan

ARMS (2):
- BIBR 277 tablet (Experimental)
  Interventions: Drug: BIBR 277 tablet
- BIBR 277 capsule (Active Comparator)
  Interventions: Drug: BIBR 277 capsule

INTERVENTIONS:
Drug: BIBR 277 tablet
  Other Names: Telmisartan
  Arms: BIBR 277 tablet
Drug: BIBR 277 capsule
  Other Names: Telmisartan
  Arms: BIBR 277 capsule

SUMMARY:
Study to investigate the bioequivalence of BIBR 277 tablet (Erythritol based) vs. BIBR 277 capsule

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 20 and <= 35 years
2. Weight: BMI >= 17.6 and <= 26.4 (Weight (kg) / Height (m)2)
3. Subjects judged by the investigator to be eligible as study subjects, with no clinically significant findings after screening
4. Subjects who volunteer to participate and are able to fully understand and agree with this study by written informed consent

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
3. Chronic or relevant acute infections
4. History of hepatic disorder (e.g., biliary cirrhosis, cholestasis)
5. History of serious renal disorder
6. History of or present bilateral renal artery stenosis or lack of unilateral kidney accompanying arterial stenosis
7. History of or present cerebrovascular disorder
8. History of hyperkalemia
9. History of hypersensitivity to active ingredient (Telmisartan) or other angiotensin II receptor antagonists
10. History of or present orthostatic hypotension or faint
11. Surgery of gastrointestinal tract (except appendectomy)
12. History of alcohol or drug abuse
13. Participation to another trial with an investigational drug within 4 months prior to the trial
14. Whole blood donation more than 400 mL within 3 months prior to the trial
15. Whole blood donation more than 100 mL within 1 month prior to the trial
16. Donation of constituent of blood of more than 400 mL within 1 month prior to the trial
17. Any medication which might influence the result of the trial within 10 days prior to the trial
18. Excessive physical activities within 7 days prior to the trial
19. Alcohol drinking within 3 days prior to the trial
20. Inability to comply with restriction of protocol
21. Other than above, those who are judged by the investigator to be inappropriate as the subjects of the study

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2002-07; Primary Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum observed concentration of the Telmisartan in plasma) | up to 72 hours after drug administration
AUC0-72hr (area under the concentration-time curve of the Telmisartan in plasma from zero time to 72hr | up to 72 hours after drug administration

SECONDARY OUTCOMES:
Individual time courses of the Telmisartan plasma concentrations | up to 72 hours after drug administration
tmax (time to reach Cmax) | up to 72 hours after drug administration
t1/2 (terminal half-life of the Telmisartan in plasma) | up to 72 hours after drug administration
AUC0-∞(area under the concentration-time curve of Telmisartan in plasma from zero time to infinity) | up to 72 hours after drug administration
MRT0-∞ (total mean residence time of Telmisartan molecules in the body) | up to 72 hours after drug administration
Number of subjects with adverse events | up to 72 hours after last drug administration
Number of subjects with clinically significant findings in vital signs | up to 72 hours after last drug administration
  blood pressure, pulse rate
Number of subjects with clinically significant findings in laboratory tests | up to 72 hours after last drug administration
Number of subjects with clinically significant findings in ECG | up to 72 hours after last drug administration